CLINICAL TRIAL: NCT06908356
Title: An Open Label Clinical Trial to Evaluate the Efficacy and Safety of PRAX-628 in Adult Patients With Focal Onset or Primary Generalized Tonic-Clonic Seizures
Brief Title: An Open Label Trial to Evaluate the Efficacy and Safety of PRAX-628 in Adults With Focal Onset or Tonic-Clonic Seizures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRAX-628-212
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Focal Onset Seizure; Primary Generalized Epilepsy
Keywords: Focal Onset Seizure; Primary Generalized Epilepsy; Tonic-Clonic
MeSH Terms: conditions — Seizures; Epilepsy, Idiopathic Generalized

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label 30mg/day PRAX-628 for 8 weeks (Experimental): Participants who meet all eligibility criteria will receive 30mg of PRAX-628 for 8 weeks.
  Interventions: Drug: 30mg PRAX-628

INTERVENTIONS:
Drug: 30mg PRAX-628 — Once daily oral

SUMMARY:
An Open Label Clinical Trial to Evaluate the Efficacy and Safety of PRAX-628 in Adult Patients With Focal Onset or Primary Generalized Tonic-Clonic Seizures

DETAILED DESCRIPTION:
An open label clinical trial to evaluate the efficacy and safety of PRAX-628 in adult patients with focal onset or primary generalized tonic-clonic seizures who can attest to concurrently taking at least 1, but no more than 3 acceptable anti-seizure medications.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of focal onset seizures or idiopathic generalized tonic clonic seizures.
* Evidence by computed tomography (CT) or magnetic resonance imaging (MRI) in the past that has ruled out a progressive cause of epilepsy.
* Participant must have been receiving stable doses of allowable ASMs (a minimum of 1 and a maximum of 3 ASMs).
* Participant and/or caregiver (if applicable) self-reports at least 2 countable focal onset seizures per month for focal onset patients, or 1 countable generalized tonic-clonic seizure per month in the 3 months immediately prior to the Screening/Observation Period for PGTCS patients.

Exclusion Criteria:

* History of pseudo or psychogenic seizures, or cluster seizures only, within the 12-month period preceding study entry where the individual seizures cannot be counted, or an episode of convulsive status epilepticus requiring hospitalization and intubation in the 12 months prior to Screening.
* Planned epilepsy surgery during the course of the clinical trial.
* History of neurosurgery for seizures <1 year prior to enrollment, or radiosurgery <2 years prior to enrollment.
* Schizophrenia and obsessive-compulsive disorder, or other serious mental health disorders.
* Active suicidal plan/intent in the past 6 months, or a history of suicide attempt in the last 2 years, or more than 1 lifetime suicide attempt.
* Participants with a history of malignancy, myeloproliferative or lymphoproliferative disorders within the past 5 years are excluded.
* History of cardiac disease(s)/cardiac conduction disorders/or cardiac structural abnormality(ies).
* Is pregnant or breastfeeding at the time of Screening, or has a positive serum pregnancy test at Screening or is planning to become pregnant during the clinical trial or within 14 days of the last study drug dose.
* Has received any other experimental or investigational drug, device or other therapy within 30 days or 5 half-lives (whichever is longer) prior to Screening, or any prior use of gene therapy.
* Vigabatrin: Use in the last 5 years without stable visual fields tested twice over the 12 months after the last dose of vigabatrin.
* Felbamate: If used as a concomitant ASM, patients must be on felbamate for at least 2 years, with a stable dose for 2 months prior to Screening. If a patient received felbamate in the past, it must have been discontinued 2 months prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of PRAX-628 on seizure frequency in adults with FOS or PGTCS currently taking ASMs | 8 weeks
  Median percent change in monthly (28 days) seizure frequency from the Screening/Observation Period to the Treatment Period for PRAX-628

SECONDARY OUTCOMES:
To evaluate the efficacy of PRAX 628 on seizure frequency in adults with FOS or PGTCS currently taking ASMs | 8 weeks
  • Proportion of participants experiencing a ≥50% reduction in monthly (28 days) seizure frequency from the Screening/Observation Period to the Treatment Period (Responder Rate) for PRAX-628.
To evaluate the efficacy of PRAX 628 on seizure frequency in adults with FOS or PGTCS currently taking ASMs | 8 weeks
  • Proportion of participants experiencing seizure freedom, 100% reduction in monthly (28 days) seizure frequency from the Screening/Observation Period to the Treatment Period for PRAX-628.
To evaluate the efficacy of PRAX 628 on seizure frequency in adults with FOS or PGTCS currently taking ASMs | 8 weeks
  • Number of days after the first administration of PRAX-628 to reach the same or higher number of monthly seizures from the Screening/Observation Period to the Treatment Period
CGI-S Change from Baseline | 8 weeks
  CGI-S assesses the clinician's impression of the participant's current illness state. The clinician should use his/her total clinical experience with this patient population and rate the current severity on a 7-point scale from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
PGI-S Change from Baseline | 8 weeks
  PGI-S assesses the participants' impression of their current illness state. The participant is required to assess their condition on a 7-point scale from 1 (Not present) to 7 (extremely severe).
To assess the safety and tolerability of PRAX-628 in adults with FOS or PGTCS currently taking ASMs | 8 weeks
  The number of participants with Adverse Events (AE) will be reported by preferred term

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Praxis Precision Medicines
Locations (11):
- United States (8):
  - Praxis Research Site, Phoenix, Arizona
  - Praxis Research Site, Miami Lakes, Florida
  - Praxis Research Site, Bethesda, Maryland
  - Praxis Research Site, Chesterfield, Missouri
  - Praxis Research Site, Hackensack, New Jersey
  - Praxis Research Site, Middletown, New York
  - Praxis Research Site, Round Rock, Texas
  - Praxis Research Site, Seabrook, Texas
- Australia (2):
  - Praxis Research Site, Heidelberg
  - Praxis Research Site, Melbourne
- Praxis Research Site, Madrid, Spain